CLINICAL TRIAL: NCT01248637
Title: A Clinical Trial of Intratumoral Hypoxia and Its Biologic Correlates in Patients Undergoing Surgical Resection of Localized Pancreatic Cancer, Using Pre-operative Administration of the Hypoxia Marker Pimonidazole.
Brief Title: Study of Intratumoral Hypoxia Using Pre-operative Administration of Pimonidazole
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: PIMO-PANC; UHN REB 10-0350-C
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; pancreatic cancer; pancreatic tumor; pimonidazole; hypoxia; whipple's resection
MeSH Terms: conditions — Pancreatic Neoplasms; Hypoxia | interventions — pimonidazole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Pancreatic Tumor biopsy and blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pimonidazole hydrochloride: Oral pimonidazole is administered at a dose of 0.5gm/m2 once approximately 24 hrs prior to surgery
  Interventions: Drug: Pimonidazole hydrochloride

INTERVENTIONS:
Drug: Pimonidazole hydrochloride — Pimonidazole is a 2-nitroimidazole that is selectively reduced and covalently binds to intracellular macromolecules in areas of hypoxia (by definition, p02 <= 10mm Hg) within normal and tumour tissue. Pimonidazole adducts can then be detected by immunolabelling techniques (microscopy, ELISA, flow cytometry etc). In this study, pimonidazole will be administered orally as a one time dose of 0.5gm/m2 24hrs prior to surgery. Since the drug has a half-life of approximately 5 hrs, this time-frame ensures low circulating levels at the time of surgery and therefore reduces the confounding effects of surgical hypoxia on tumour analysis.
  Other Names: Hypoxyprobe-1

SUMMARY:
This study involves the administration of a hypoxia marker, pimonidazole hydrochloride, taken orally approximately 24 hours before surgical resection of a pancreatic tumor in order to identify areas of lower oxygen content on tumor samples.

DETAILED DESCRIPTION:
Intratumoral hypoxia (low oxygen concentration or pO2) occurs when oxygen consumption exceeds its delivery by the vascular system. Hypoxia is associated with adverse patient outcome in many human cancers and this association is hypothesized to be due to a combination of treatment resistance and aggressive tumor biology.

The study of hypoxia is also important as new cancer drugs are being developed that are specifically active on cancer cells in area of tumors with lower oxygen levels.

his study involves administering the hypoxia probe pimonidazole hydrochloride to patients prior to resection of pancreatic adenocarcinoma to evaluate the extent, molecular context and clinical relevance of hypoxia in clinical pancreatic cancer samples and the subsequently derived primary xenograft tumors.

We propose accrual of patients over a 5-year period to evaluate hypoxia within 100 clinical tumor specimens and corresponding primary xenograft tumours where available. The complementary techniques of wide-field multicolor fluorescence image analysis microscopy and high level flow cytometry will be used to identify potential relationships between intratumoral hypoxia and cell proliferation, differentiation, and the expression of putative cancer stem cell markers.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* provisional diagnosis of pancreatic cancer
* scheduled resection at UHN
* consented to ICGC Pancreatic Cancer Genome Project
* surgery planned for >2 days away (drug administration has to be 16-20hrs before surgery)

Exclusion Criteria:

* not participating in ICGC
* contraindications to pimonidazole (allergy)
* surgery scheduled for same or next day (not enough time to arrange for drug administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating in ICGC Pancreatic Cancer Genome Project.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
characterization of intratumoral hypoxia in pancreatic cancer | 5 Years
  estimation of tumoral hypoxic fraction by immunodetection of pimonidazole adducts.
correlation of intratumoral hypoxia with patient survival rate | 5 Years
  evaluation of correlation of tumoral hypoxia with disease-free survival using Cox proportional hazards analysis

SECONDARY OUTCOMES:
correlation of hypoxia with molecular markers | 5 Years
  colocalization of molecular markers using immunofluorescence microscopy: Stem-cell like populations markers of EMT Endogenous markers of hypoxia (HIF1a, CAIX)
to assess utility of circulating osteopontin and miR-210 for identifying hypoxia | 5 Years
  correlation of tumoral hypoxic fraction with plasma levels of osteopontin and miR-210

CONTACTS AND LOCATIONS:
Overall Officials: Neesha Dhani, MD, Principal Investigator — Univeristy Health Network - Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dhani NC, Serra S, Pintilie M, Schwock J, Xu J, Gallinger S, Hill RP, Hedley DW. Analysis of the intra- and intertumoral heterogeneity of hypoxia in pancreatic cancer patients receiving the nitroimidazole tracer pimonidazole. Br J Cancer. 2015 Sep 15;113(6):864-71. doi: 10.1038/bjc.2015.284. Epub 2015 Sep 1. PMID 26325106